CLINICAL TRIAL: NCT02696031
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study of Secukinumab 150 mg in Patients With Active nr- axSpA to Evaluate the Safety,Tolerability and Efficacy up to 2 Yrs, Followed by an Opt Phase of Either 150 mg or 300 mg Randomized Dose Escalation for up to Another 2 Yrs
Brief Title: Study of Efficacy and Safety of Secukinumab in Patients With Non-radiographic Axial Spondyloarthritis
Acronym: PREVENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457H2315
Record Dates: First submitted 2015-10-13; First posted 2016-03-02 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Non-radiographic Spondyloarthritis
Keywords: non-radiographic spondyloarthritis; axial spondyloarthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: This was a randomized, double-blind, placebo-controlled study. Approximately 555 patients were randomized to one of three treatment groups (secukinumab 150 mg Load, secukinumab 150 mg No Load or placebo in a ratio of 1:1:1):
  * Group 1 (secukinumab 150 mg Load): secukinumab 150 mg (1 mL, 150 mg/mL) s.c. prefilled syringe (PFS) at baseline (BSL), Weeks 1, 2 and 3, followed by administration every four weeks starting at Week 4
  * Group 2 (secukinumab 150 mg No Load): secukinumab 150 mg (1 mL, 150 mg/mL) s.c. PFS at BSL, placebo at Weeks 1, 2 and 3, followed by secukinumab 150 mg PFS administration every four weeks starting at Week 4
  * Group 3 (placebo): placebo (1 mL) s.c. PFS at BSL, Weeks 1, 2, 3, followed by administration every four weeks starting at Week 4 Based on the clinical judgment of disease activity by the investigator and the patient, background medications, such as NSAIDs and DMARDs, may have been modified or added to treat signs and symptoms of nr-axSpA from Week 16 on.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Secukinumab, 150 mg Load (Core phase) (Experimental): Secukinumab 150 mg s.c., pre-filled syringe (PFS) at baseline, Weeks 1, 2, and 3, followed by administration every four weeks starting at Week 4, Load, Core phase
  Interventions: Drug: Secukinumab
- Secukinumab, 150 mg No Load (Core phase) (Experimental): Secukinumab 150 mg s.c. PFS at baseline, placebo at Weeks 1, 2, and 3, followed by secukinumab 150 mg PFS administration every four weeks starting at Week 4, No Load, Core phase
  Interventions: Drug: Secukinumab
- Placebo (Core phase) (Placebo Comparator): Placebo s.c., PFS at baseline, Weeks 1, 2, 3, followed by administration every four weeks starting at Week 4, Core phase
  Interventions: Drug: Placebo
- Core Phase Responder 150 mg (Extension phase) (Experimental): Core Phase Responder 150 mg blinded: secukinumab 150 mg s.c. PFS and placebo (1 mL) s.c. PFS every four weeks, in the Extension phase
  Interventions: Drug: Secukinumab; Drug: Placebo
- Core Phase Responder 300 mg (Extension phase) (Experimental): Core Phase Responder 300 mg blinded: 2 injections with secukinumab 150 mg s.c. PFS every four weeks, in the Extension phase
  Interventions: Drug: Secukinumab
- Core Phase Non-Responder 300 mg (Extension phase) (Experimental): Core Phase Non-Responder 300 mg: 2 injections with secukinumab 150 mg s.c. PFS every four weeks open-label, in the Extension phase
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Induction: 4x 150 mg Secukinumab s.c. weekly Maintenance: 150 mg Secukinumab s.c. monthly
  Other Names: AIN457
  Arms: Core Phase Non-Responder 300 mg (Extension phase); Core Phase Responder 150 mg (Extension phase); Core Phase Responder 300 mg (Extension phase); Secukinumab, 150 mg Load (Core phase); Secukinumab, 150 mg No Load (Core phase)
Drug: Placebo — Induction: 4x placebo s.c. weekly Maintenance: placebo s.c. monthly
  Other Names: AIN457
  Arms: Core Phase Responder 150 mg (Extension phase); Placebo (Core phase)

SUMMARY:
The purpose of this study was to demonstrate the clinical efficacy, safety and tolerability of secukinumab compared to placebo in patients with nr-axSpA at Week 16 as well as Week 52 and long term efficacy and safety up to Week 104 (core phase) followed by an optional extension phase consisting of a 16-week randomized dose escalation treatment period and a continuous treatment period for up to Week 208

DETAILED DESCRIPTION:
Patients were randomized to one of three treatment groups (1:1:1) in the core phase:

* Secukinumab 150 mg Load: secukinumab 150 mg (1 mL, 150 mg/mL) s.c. pre-filled syringe (PFS) at baseline, Weeks 1, 2, and 3, followed by administration every four weeks starting at Week 4
* Secukinumab 150 mg No Load: secukinumab 150 mg (1 mL, 150 mg/mL) s.c. PFS at baseline, placebo at Weeks 1, 2, and 3, followed by secukinumab 150 mg PFS administration every four weeks starting at Week 4
* Placebo: placebo (1 mL) s.c. PFS at baseline, Weeks 1, 2, 3, followed by administration every four weeks starting at Week 4.

All patients received secukinumab 150 mg as open-label treatment from Week 52 up to Week 100, unless they had discontinued study treatment.

At Week 104, all patients who finished the core phase according to the protocol were asked to continue in an optional, exploratory extension phase. Patients who achieved ASAS20 response at Week 104 (Core Phase Responders) were randomized to the following treatment groups (blinded) in the extension phase:

* Core Phase Responder 150 mg: secukinumab 150 mg (1 mL, 150 mg/mL) s.c. PFS and placebo (1 mL) s.c. PFS every four weeks;
* Core Phase Responder 300 mg: 2 injections with secukinumab 150 mg (1 mL, 150 mg/mL) s.c. PFS every four weeks.

Core Phase Non-Responders (not achieving ASAS20 at Week 104) were escalated to secukinumab 300 mg in an open-label manner.

- Core Phase Non-Responder 300 mg: 2 injections with secukinumab 150 mg (1 mL, 150 mg/mL) s.c. PFS every four weeks open-label.

Starting from Week 156 onward, a patient could switch to secukinumab 300 mg open-label based on the clinical judgment of disease activity by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female patients at least 18 years of age
* Diagnosis of axial spondyloarthritis according to Ankylosing SpondyloArthritis International Society (ASAS) axial spondyloarthritis criteria
* objective signs of inflammation (magnetic resonance imaging (MRI) or abnormal C-reactive protein)
* active axial spondyloarthritis as assessed by total Bath Ankylosing Spondylitis Disease Activity Index >=4 cm
* Spinal pain as measured by Bath Ankylosing Spondylitis Disease Activity Index question #2 ≥ 4 cm (0-10 cm) at baseline
* Total back pain as measured by Visual Analogue scale ≥ 40 mm (0-100 mm) at baseline
* Patients should have been on at least 2 different non-steroidal anti-inflammatory drugs with an inadequate response
* Patients who have been on a Tumor Necrosis Factor (TNF) α inhibitor (not more than one) must have experienced an inadequate response

Exclusion Criteria:

* Patients with radiographic evidence for sacroiliitis, grade ≥ 2 bilaterally or grade ≥ 3 unilaterally
* Inability or unwillingness to undergo MRI
* Chest X-ray or MRI with evidence of ongoing infectious or malignant process
* Patients taking high potency opioid analgesics
* Previous exposure to secukinumab or any other biologic drug directly targeting interleukin-17 (IL-17) or IL-17 receptor
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (126):
- United States (18):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Idaho Falls, Idaho
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, Lansing, Michigan
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Potsdam, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Leander, Texas
  - Novartis Investigative Site, Mesquite, Texas
- Australia (5):
  - Novartis Investigative Site, Coffs Harbour, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
  - Novartis Investigative Site, Woolloongabba
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Czechia (4):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brno-Zidonice, CZE
  - Novartis Investigative Site, Brno, CZ
  - Novartis Investigative Site, Uherské Hradiště
- France (8):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Monaco
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rouen
- Germany (10):
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Potsdam
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Veszprém
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Pisa
- Japan (6):
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
- Mexico (4):
  - Novartis Investigative Site, Torreón, Coahuila
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Culiacan, State of Mexico
  - Novartis Investigative Site, Metepec, State of Mexico
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
- Norway (2):
  - Novartis Investigative Site, Kongsvinger
  - Novartis Investigative Site, Moss
- Poland (4):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (4):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
- Russia (7):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Seoul, South Korea
- Spain (13):
  - Novartis Investigative Site, Elda, Alicante
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uppsala
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Fribourg
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- United Kingdom (9):
  - Novartis Investigative Site, Westcliff-on-Sea, Essex
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Worthing, West Sussex
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Northampton
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://clinicalstudydatarequest.com/Default.aspx

REFERENCES:
- [Derived] Jamaludin A, Windsor R, Ather S, Kadir T, Zisserman A, Braun J, Gensler LS, Ostergaard M, Poddubnyy D, Coroller T, Porter B, Ligozio G, Readie A, Machado PM. Automated detection of spinal bone marrow oedema in axial spondyloarthritis: training and validation using two large phase 3 trial datasets. Rheumatology (Oxford). 2025 Oct 1;64(10):5446-5454. doi: 10.1093/rheumatology/keaf323. PMID 40489668
- [Derived] Braun J, Blanco R, Marzo-Ortega H, Gensler LS, Van den Bosch F, Hall S, Kameda H, Poddubnyy D, van de Sande M, van der Heijde D, Zhuang T, Stefanska A, Readie A, Richards HB, Deodhar A. Two-year imaging outcomes from a phase 3 randomized trial of secukinumab in patients with non-radiographic axial spondyloarthritis. Arthritis Res Ther. 2023 May 16;25(1):80. doi: 10.1186/s13075-023-03051-5. PMID 37194094
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Braun J, Blanco R, Marzo-Ortega H, Gensler LS, van den Bosch F, Hall S, Kameda H, Poddubnyy D, van de Sande M, Wiksten AS, Porter BO, Shete A, Richards HB, Haemmerle S, Deodhar A. Secukinumab in non-radiographic axial spondyloarthritis: subgroup analysis based on key baseline characteristics from a randomized phase III study, PREVENT. Arthritis Res Ther. 2021 Sep 4;23(1):231. doi: 10.1186/s13075-021-02613-9. PMID 34481517
- [Derived] Deodhar A, Blanco R, Dokoupilova E, Hall S, Kameda H, Kivitz AJ, Poddubnyy D, van de Sande M, Wiksten AS, Porter BO, Richards HB, Haemmerle S, Braun J. Improvement of Signs and Symptoms of Nonradiographic Axial Spondyloarthritis in Patients Treated With Secukinumab: Primary Results of a Randomized, Placebo-Controlled Phase III Study. Arthritis Rheumatol. 2021 Jan;73(1):110-120. doi: 10.1002/art.41477. Epub 2020 Nov 24. PMID 32770640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1583 patients were screened for this study, of which 555 patients (35.1%) were randomized. Overall, 1028 patients (64.9%) discontinued prior to screening phase completion, most due to screen failure (1000 patients, 63.2%).
Groups:
- Secukinumab, Load, Core Phase: AIN457 150 mg s.c. load, Core Phase
- Secukinumab, No Load, Core Phase: AIN457 150 mg s.c. no load, Core Phase
- Placebo, Core Phase: Placebo s.c., Core Phase
- AIN457 150 mg Extension Phase: AIN457 150 mg Core Phase Responders who were rerandomized at week 104 to the 150 mg in the Extension phase (from Week 104 to week 208).
- AIN457 300 mg Extension Phase: AIN457 150 mg Core Phase Responders who were rerandomized at week 104 to the 300 mg in the Extension phase (from Week 104 to week 208).
- AIN457 300 mg Open Label Extension Phase: AIN457 150 mg Open Label Core Phase Non-Responders who were assigned at week 104 to the 300 mg Open Label in the Extension phase (from Week 104 to week 208).
Period: Up to Week 24
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase | AIN457 150 mg Extension Phase | AIN457 300 mg Extension Phase | AIN457 300 mg Open Label Extension Phase
Started | 185 | 184 | 186 | 0 | 0 | 0
Completed (Completed week 24) | 175 | 177 | 175 | 0 | 0 | 0
Not Completed | 10 | 7 | 11 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 5 | 0 | 0 | 0
Period: Up to Week 52
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase | AIN457 150 mg Extension Phase | AIN457 300 mg Extension Phase | AIN457 300 mg Open Label Extension Phase
Started | 185 | 184 | 186 | 0 | 0 | 0
Completed | 156 | 165 | 160 | 0 | 0 | 0
Not Completed | 29 | 19 | 26 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 7 | 11 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 3 | 9 | 0 | 0 | 0
Period: Up to Week 104
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase | AIN457 150 mg Extension Phase | AIN457 300 mg Extension Phase | AIN457 300 mg Open Label Extension Phase
Started | 185 | 184 | 186 | 0 | 0 | 0
Completed | 146 | 143 | 149 | 0 | 0 | 0
Not Completed | 39 | 41 | 37 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 10 | 16 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 12 | 11 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 11 | 5 | 0 | 0 | 0
Not completed — Pt completed wk 52. Withdrawal by subject at wk 52. | 0 | 1 | 0 | 0 | 0 | 0
Period: Extension Phase From wk 104 to wk 208
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase | AIN457 150 mg Extension Phase | AIN457 300 mg Extension Phase | AIN457 300 mg Open Label Extension Phase
Started | 0 | 0 | 0 | 147 | 147 | 78
Completed | 0 | 0 | 0 | 137 | 132 | 72
Not Completed | 0 | 0 | 0 | 10 | 15 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6 | 8 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase | Total
Number analyzed (Participants) | 185 | 184 | 186 | 555
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 183 | 180 | 183 | 546
  >=65 years | 2 | 4 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (11.45) | 39.8 (11.68) | 39.3 (11.47) | 39.4 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 100 | 95 | 300
  Male | 80 | 84 | 91 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 7 | 24
  Not Hispanic or Latino | 165 | 162 | 161 | 488
  Unknown or Not Reported | 11 | 14 | 18 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 4 | 8 | 11 | 23
  Black or African American | 0 | 2 | 1 | 3
  White | 176 | 165 | 167 | 508
  Other | 5 | 7 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of TNF Naive Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 40 Response at Week 16
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the VAS signifies higher severity.
Time Frame: Week 16
Population: Subset of TNF naive patients
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 164 | 166 | 171
Participants | 68 | 70 | 50
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0197, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.09 to 2.70]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0146, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.12 to 2.76]

2. Primary Outcome: The Number and Percentage of TNF Naive Participants Who Achieved an Assessment of SpondyloArthritis International Society (ASAS) 40 Response at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: Subset of TNF naive patients
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 164 | 166 | 171
Participants | 58 | 66 | 34
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 52; Test type: Superiority; p = 0.0017, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.35 to 3.63]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 52; Test type: Superiority; p < .0001, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.64 to 4.36]

3. Secondary Outcome: The Number and Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society (ASAS) 40 Response
Description: as for outcome 1
Time Frame: Week 16 and week 52
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 185 | 184 | 186
Participants
  week 16 | 74 | 75 | 52
  week 52 | 62 | 70 | 36
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0108, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.14 to 2.74]; Odds ratio, 95% CI, and p-value were from a logistic regression model with treatment, stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNFi status as factors and baseline weight as a covariate
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0087, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.16 to 2.78]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; Test type: Superiority — week 52; p = 0.0016, Regression, Linear — unadjusted p-value; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.34 to 3.49]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; Test type: Superiority — week 52; p < .0001, Regression, Linear — unadjusted p-value; Median Difference (Net) = 2.61, 95% CI 2-sided [1.62 to 4.19]; [other analysis details as in outcome 3, analysis 1]

4. Secondary Outcome: The Number and Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society (ASAS) 20 Response
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS 20 response is defined as an improvement of ≥20% and ≥1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain. A higher score on the VAS signifies higher severity.
Time Frame: Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 185 | 184 | 186
Participants | 105 | 107 | 85
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0260, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.06 to 2.43]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0149, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.11 to 2.54]; [other analysis details as in outcome 3, analysis 1]

5. Secondary Outcome: The Number and Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society (ASAS) 5/6 Response
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  The ASAS 5/6 improvement criteria is an improvement of ≥20% in at least five of all six domains. A higher score on the VAS signifies higher severity.
Time Frame: Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 185 | 184 | 186
Participants | 74 | 66 | 44
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0005, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.43 to 3.58]; Odds ratio, 95% CI, and p-value were from a logistic regression model with treatment, stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNF-alpha status as factors and baseline weight as a covariate
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0094, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.16 to 2.94]; [other analysis details as in outcome 5, analysis 1]

6. Secondary Outcome: The Number and Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society Partial Remission (ASAS PR)
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  The ASAS partial remission criteria are defined as a value not above 2 units in each of the four main domains on a scale of 10. A higher score on the VAS signifies higher severity.
Time Frame: Week 16
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 185 | 184 | 186
Participants | 40 | 39 | 13
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p < .0001, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 3.80, 95% CI 2-sided [1.95 to 7.39]; [other analysis details as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0001, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 3.64, 95% CI 2-sided [1.87 to 7.10]; [other analysis details as in outcome 5, analysis 1]

7. Secondary Outcome: Change in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) is a set of 10 questions designed to determine the degree of functional limitation in those subjects with AS. The ten questions were chosen with a major input from subjects with AS. The first 8 questions consider activities related to functional anatomy. The final 2 questions assess the subjects' ability to cope with everyday life. A 100 mm visual analog scale (VAS) is used to answer the questions. The mean of the ten questions gives the BASFI score - a value between 0 and 10. (0 being no problem and 10 being the worst problem, captured as a continuous visual analog scale (VAS)). A higher score on the VAS signifies higher severity.
Time Frame: Baseline and Week 16
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 181 | 177 | 177
Index | -1.75 (0.202) | -1.64 (0.204) | -1.01 (0.206)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0041, MMRM — unadjusted p-value; LS Mean = -0.75, 95% CI 2-sided [-1.26 to -0.24], Standard Error of Mean 0.259; LS Mean, 95% CI, and p-value were from a mixed model repeated measures (MMRM) with treatment group, analysis visit, stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNFi status as factors, weight and baseline score as covariates, treatment by analysis visit and baseline score by analysis visit as interaction terms, using an unstructured covariance structure
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0143, MMRM — unadjusted p-value; LS Mean = -0.64, 95% CI 2-sided [-1.15 to -0.13], Standard Error of Mean 0.259; [other analysis details as in outcome 7, analysis 1]

8. Secondary Outcome: The Number and Percentage of Patients to Achieve a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response
Description: The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) consists of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which is used to answer 6 questions pertaining to the 5 major symptoms of AS. The BASDAI 50 is defined as an improvement of at least 50% in the BASDAI compared to baseline. A higher score on the VAS signifies higher severity.
Time Frame: Week 16 and 52
Population: Full Analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 185 | 184 | 186
Participants
  week 16 | 69 | 69 | 39
  week 52 | 57 | 65 | 37
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0001, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.58 to 4.07]; Odds ratio, 95% CI, and p-value were from a logistic regression model with treatment, stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNFi status as factors and baseline weight and baseline score as covariates. Missing responses for any reason were imputed as non-responders
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0002, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.51 to 3.89]; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 52; Test type: Superiority; p = 0.0056, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.22 to 3.24]; [other analysis details as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 52; Test type: Superiority; p = 0.0005, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.45 to 3.78]; [other analysis details as in outcome 8, analysis 1]

9. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a validated assessment tool using 1 through 10 scales (1 indicating "no problem" and 10 indicating " worst problem"), to characterize six clinical domains (fatigue, spinal pain, joint pain/selling, localized tenderness, morning stiffness duration, morning stiffness severity) pertaining to five major symptoms of Ankylosing Spondylitis (AS). The computed final BASDAI score is a value between 0 and 10 with a higher score indicating worse disease. A higher score on the VAS signifies higher severity.
Time Frame: Baseline and Week 16
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 181 | 177 | 177
scores on a scale | -2.35 (0.201) | -2.43 (0.203) | -1.46 (0.205)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0006, mixed model repeated measures (MMRM) — unadjusted p-value; LS Mean of treatment difference = -0.89, 95% CI 2-sided [-1.39 to -0.38], Standard Error of Mean 0.256; [other analysis details as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0002, mixed model repeated measures (MMRM) — unadjusted p-value; LS Mean of Treatment Difference = -0.97, 95% CI 2-sided [-1.47 to -0.47], Standard Error of Mean 0.255; [other analysis details as in outcome 7, analysis 1]

10. Secondary Outcome: Change in Ankylosing Spondylitis Quality of Life (ASQoL) Scores at Week 16
Description: The Ankylosing Spondylitis Quality of Life scores (ASQoL) is a self-administered questionnaire designed to assess health-related quality of life in adult patients with Ankylosing Spondylitis. The ASQoL contains 18 items with a dichotomous yes/no response option. A single point is assigned for each "yes" response and no points for each "no" response resulting in overall scores that range from 0 (least severity) to 18 (highest severity). As such, lower score indicate better quality of life. Items include an assessment of mobility/energy, self-care and mood/emotion. The recall period is "at the moment," and the measure requires approximately 6 minutes to complete.
Time Frame: Baseline and Week 16
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 181 | 176 | 177
Scores on a scale | -3.45 (0.408) | -3.62 (0.414) | -1.84 (0.421)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0008, MMRM — unadjusted p-value; LS Mean = -1.61, 95% CI 2-sided [-2.54 to -0.67], Standard Error of Mean 0.478; LS Mean, 95% CI, and p-value are from a mixed model repeated measures (MMRM) with treatment group, analysis visit, stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNFi status as factors, weight and baseline score as covariates, treatment by analysis visit and baseline score by analysis visit as interaction terms, using an unstructured covariance structure
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0002, MMRM — unadjusted p-value; LS Mean = -1.78, 95% CI 2-sided [-2.72 to -0.84], Standard Error of Mean 0.479; [other analysis details as in outcome 10, analysis 1]

11. Secondary Outcome: Change in Ankylosing Spondylitis Quality of Life (ASQoL) Scores at Week 52
Description: The Ankylosing Spondylitis Quality of Life scores (ASQoL) is a self-administered questionnaire designed to assess health-related quality of life in adult patients with Ankylosing Spondylitis. The ASQoL contains 18 items with a dichotomous yes/no response option. A single point is assigned for each "yes" response and no points for each "no" response resulting in overall scores that range from 0 (least severity) to 18 (highest severity). As such, lower score indicate better quality of life. Items include an assessment of mobility/energy, self-care and mood/emotion. The recall period is "at the moment," and the measure requires approximately 6 minutes to complete.
  Summary statistics are presented for participants (n) without intercurrent events.
Time Frame: Baseline and Week 52
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 83 | 88 | 54
Scores on a scale | -7.1 (4.77) | -7.6 (5.38) | -6.4 (4.64)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; Test type: Superiority; p = 0.0012, Wilcoxon (Mann-Whitney) — unadjusted p-value; The endpoint was analyzed by composite estimand strategy. Extreme unfavorable value is assigned for patients with treatment escape or missing data
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; Test type: Superiority; p < .0001, Wilcoxon (Mann-Whitney) — unadjusted p-value; [statistical method as in outcome 11, analysis 1]

12. Secondary Outcome: The Number and Percentage of Patients Who Achieved an Ankylosing Spondylitis Disease Activity Score (ASDAS)-C-Reactive Protein (CRP) Inactive Disease
Description: Ankylosing Spondylitis Disease Activity Score (ASDAS) - C-reactive protein (CRP) inactive disease criteria are defined as a value below 1.3. Higher score indicates worse symptoms. The formula is: ASDAS-CRP = 0.121 x total back pain + 0.110 x patient global + 0.073 x peripheral pain/swelling + 0.058 x duration of morning stiffness + 0.579 x ln(hsCRP +1)
Time Frame: Week 52
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 185 | 184 | 186
Participants | 29 | 44 | 19
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 52; Test type: Superiority; p = 0.0577, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.98 to 3.45]; Odds ratio, 95% CI, and p-value were from a logistic regression model with treatment, stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNFi status as factors and baseline weight and baseline score as covariates. Missing responses for any reason were imputed as non-responders. Patients were considered as non-responders after treatment switch decision
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 52; Test type: Superiority; p = 0.0003, Regression, Logistic — unadjusted p-value; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.65 to 5.41]; [other analysis details as in outcome 12, analysis 1]

13. Secondary Outcome: Change in High Sensitivity C-reactive Protein
Description: High sensitivity C-reactive protein is measured as a marker of inflammation from blood samples during the study.
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 180 | 176 | 175
ratio | 0.64 (1.078) | 0.64 (1.079) | 0.91 (1.080)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0002, MMRM — unadjusted p-value; Relative Treatment Effect = 0.70, 95% CI 2-sided [0.58 to 0.84]; Analysis was done on the log(e) ratio of the treatment value vs. baseline value to normalize the distribution of the hsCRP at each visit. LS Mean, SE, 95% CI and p-value were from mixed-effect model repeated measures (MMRM) with treatment, visit, stratification factor and TNFi status as factors, log(e) baseline and weight as covariates, treatment by visit and log(e) baseline by visit as interaction terms and an unstructured covariance
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0002, MMRM — unadjusted p-value; Relative Treatment Effect = 0.70, 95% CI [0.58 to 0.84]; Analysis was done on the log(e) ratio of the treatment value vs. baseline value to normalize the distribution of the hsCRP at each visit. LS Mean, SE, 95% CI and p-value were from mixed-effect model repeated measures (MMRM) with treatment, visit, stratification factor and TNFi status as factors, log(e) baseline and weight as covariates, treatment by visit and log(e) baseline by visit as interaction terms and an unstructured covariance structure

14. Secondary Outcome: Change in Short Form-36 Physical Component Summary (SF-36 PCS)
Description: The Short Form-36 Physical Component Summary (SF-36 PCS) is an instrument to measure health-related quality of life among healthy patients and patients with acute and chronic conditions.
  It consists of eight subscales (domains) that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role- Emotional, and Mental Health. Two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) also can be computed. The eight domains are based on a scale from 0-100 while PCS and MCS are norm-based scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate a higher level of functioning. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 182 | 176 | 178
Scores on a Scale | 5.71 (0.683) | 5.57 (0.694) | 2.93 (0.705)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0006, ANCOVA — unadjusted p-value; LS Mean of Treatment Difference = 2.77, 95% CI 2-sided [1.20 to 4.34], Standard Error of Mean 0.799; [other analysis details as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p = 0.0011, ANCOVA — unadjusted p-value; LS Mean of Treatment Difference = 2.64, 95% CI 2-sided [1.06 to 4.22], Standard Error of Mean 0.803; [other analysis details as in outcome 7, analysis 1]

15. Secondary Outcome: Change in Sacroiliac Joint Edema - Week 16
Description: Magnetic Resonance Images (MRI) of the Sacroiliac Joint (SIJ) were assessed for the presence and severity of SIJ bone marrow edema according to the Berlin Active Inflammatory Lesions Scoring with a maximum score of 24.
Time Frame: Baseline and Week 16
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 180 | 177 | 174
Scores on a Scale | -1.68 (0.24) | -1.03 (0.18) | -0.39 (0.15)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p < 0.0001, ANCOVA — unadjusted p-value; LS Mean, 95% CI, and p-value were from an ANCOVA model with treatment group and stratification factor (CRP+/MRI+, CRP+/MRI-, CRP-/MRI+) and TNFi status as factors, weight and baseline score as covariates. Missing data were imputed using multiple imputation (MI, MAR assumption) prior to running ANCOVA
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; week 16; Test type: Superiority; p < 0.0001, ANCOVA — unadjusted p-value; [other analysis details as in outcome 15, analysis 1]

16. Secondary Outcome: Change in Sacroiliac Joint Edema - Week 52
Description: as for outcome 15
Time Frame: Baseline and Week 52
Population: Full Analysis Set where intercurrent event = no.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab, Load, Core Phase | Secukinumab, No Load, Core Phase | Placebo, Core Phase
Number analyzed (Participants) | 81 | 87 | 53
Scores on a scale | -2.9 (4.54) | -1.9 (3.40) | -0.1 (1.97)
Statistical Analysis 1: Comparison: Secukinumab, Load, Core Phase vs Placebo, Core Phase; Test type: Superiority; p < .0001, Wilcoxon (Mann-Whitney) — unadjusted p-value; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Secukinumab, No Load, Core Phase vs Placebo, Core Phase; Test type: Superiority; p < .0001, Wilcoxon (Mann-Whitney) — unadjusted p-value; [statistical method as in outcome 11, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 12 wks post-treatment, up to a maximum timeframe of 1520 days (approx. 4.2 years). Safety results summarize long term data for all patients for the entire period of their study participation, which, for the majority of pts, combines the core phase and the extension phase (not all pts participated in the extension). The table is presented by dose group, AIN457 150 mg and AIN457 300 mg and placebo.
Description: Any exposure to AIN457 in the core phase is presented as Any AIN457 150 mg, regardless if patients were initially assigned to Load or No Load. Considering the total length of exposure to AIN457 150 mg, the effect of initial loading regimen during the first 4 weeks of treatment is considered negligible.
  Pts. may have switched from placebo to 150 mg or from 150 mg to 300 mg during the course of the study. Therefore, some pts are counted in more than 1 dose group, depending on the AE timing.
Groups:
- Any AIN457 150 mg, in Core Phase and Extension Phase: Includes patients originally randomized to AIN457 150 mg (Load and No Load) at baseline and placebo patients switched to AIN457 150 mg before or at W52 (AEs occurring after the switch) who either were re-randomized (Core Phase Responders) to AIN457 150 mg at W104 or did not participate in the Extension Phase.
- Any AIN457 300 mg in Extension Phase: Includes patients re-randomized (Core Phase Responders) or re-assigned (Core Phase Non-Responders) to AIN457 300 mg at W104 (Extension Phase) and patients re-randomized (Core Phase Responders) to AIN457 150 mg at W104 who up-titrated to AIN457 300 mg (only AEs occurring after up-titration).
- Any AIN457, In Core Phase and Extension Phase: Includes patients randomized or switched (AEs occurring after the switch) to AIN457 150 mg (Load and No Load) who either were re-randomized (Core Phase Responders) to AIN457 150 mg or AIN457 300 mg at W104 or did not participate in the Extension Phase.
- Placebo, Core Phase: Includes patients originally randomized to Placebo (AEs until the time of a switch to AIN457 150 mg)
Arm/Group | Any AIN457 150 mg, in Core Phase and Extension Phase | Any AIN457 300 mg in Extension Phase | Any AIN457, In Core Phase and Extension Phase | Placebo, Core Phase
All-Cause Mortality (participants affected / at risk) | 0/543 | 0/254 | 0/543 | 0/186
Serious Adverse Events (participants affected / at risk) | 48/543 | 11/254 | 58/543 | 8/186
Other Adverse Events (participants affected / at risk) | 320/543 | 74/254 | 335/543 | 67/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg, in Core Phase and Extension Phase (N=543) | Any AIN457 300 mg in Extension Phase (N=254) | Any AIN457, In Core Phase and Extension Phase (N=543) | Placebo, Core Phase (N=186)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 3 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Vaccination site cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Viral tracheitis (Infections and infestations) | 0 | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Arthroscopy (Investigations) | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Substance-induced mood disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cervix enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Varicocele (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg, in Core Phase and Extension Phase (N=543) | Any AIN457 300 mg in Extension Phase (N=254) | Any AIN457, In Core Phase and Extension Phase (N=543) | Placebo, Core Phase (N=186)
Diarrhoea (Gastrointestinal disorders) | 55 | 6 | 61 | 10
Bronchitis (Infections and infestations) | 23 | 6 | 28 | 2
Nasopharyngitis (Infections and infestations) | 137 | 33 | 146 | 32
Pharyngitis (Infections and infestations) | 27 | 5 | 31 | 1
Sinusitis (Infections and infestations) | 30 | 5 | 34 | 3
Upper respiratory tract infection (Infections and infestations) | 65 | 16 | 77 | 13
Urinary tract infection (Infections and infestations) | 38 | 9 | 42 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 6 | 48 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 3 | 38 | 3
Headache (Nervous system disorders) | 61 | 7 | 65 | 9
Hypertension (Vascular disorders) | 29 | 5 | 34 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Publications from a single-site are postponed until publication of the pooled clinical trial data (i.e., data from all sites) or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02696031/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT02696031/SAP_002.pdf